CLINICAL TRIAL: NCT01687153
Title: Effects of Traumatic Brain Injury and Post Traumatic Stress Disorder on Alzheimer's Disease (AD) in Veterans Using Alzheimer's Disease Neuroimaging Initiative (ADNI)
Brief Title: A Study of Brain Aging in Vietnam War Veterans
Acronym: DOD-ADNI
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Telemedicine & Advanced Technology Research Center (Other); Northern California Institute of Research and Education (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul Aisen, Professor, University of Southern California
Other Study IDs: ADC-044; W81XWH-12-2-0012 (Other Grant/Funding Number: Department of Defense); W81XWH-13-1-0259 (Other Grant/Funding Number: Department of Defense); W81XWH-14-1-0462 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2012-08-31; First posted 2012-09-18 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Traumatic Brain Injury; Post Traumatic Stress Disorder; Alzheimer's Disease; Mild Cognitive Impairment
Keywords: traumatic brain injury (TBI); post traumatic stress disorder (PTSD); Alzheimer's disease (AD); mild cognitive impairment (MCI); dementia; biomarkers; amyloid; neuroimaging; cognition disorder; tau
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Alzheimer Disease; Cognitive Dysfunction; Dementia; Cognition Disorders; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, cerobrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Traumatic Brain Injury (TBI): 65-100 Vietnam Veterans with Traumatic Brain Injury (TBI), but without PTSD, mild cognitive impairment (MCI)/dementia
- Post Traumatic Stress Disorder (PTSD): 65-100 Vietnam Veterans with PTSD, but without TBI, MCI/dementia
- Controls: 65-100 Vietnam Veteran Controls without TBI or PTSD and comparable in age, gender, and education to the other cohorts
- TBI w/ MCI: 65-100 Vietnam Veterans with TBI but without PTSD who meet the criteria for MCI but not dementia
- PTSD w/ MCI: 65-100 Vietnam Veterans with PTSD but without TBI who meet the criteria for MCI but not dementia
- Controls w/ MCI: 65-100 Vietnam Veteran Controls without TBI or PTSD who meet the criteria for MCI but not dementia, and are comparable in age, gender, and education to the other cohorts

SUMMARY:
Traumatic brain injury (TBI) and post traumatic stress disorder (PTSD) are common combat related problems and may be associated with a greater risk of Alzheimer's disease (AD). The purpose of this study is to examine the possible connections between TBI and PTSD, and the signs and symptoms of AD on Veterans as they age.

The information collected will help to learn more about how these injuries may affect Veterans of the Vietnam War as they grow older, as well as Veterans of the current wars in Iraq and Afghanistan, who also have these types of combat related injuries.

DETAILED DESCRIPTION:
The overall long-term goal of this project is to prevent AD, which affects almost 50% of the US population over 85 years of age, and is the most common cause of dementia. Clinical signs and symptoms of AD include cognitive impairments, especially memory and emotional disturbances. In order to accomplish this goal of prevention, a population at risk must be identified. Evidence suggests that both TBI and PTSD increase risk for cognitive decline, AD, and dementia.

TBI and PTSD are common problems resulting from military service. Thus far, there have been no prospective studies using imaging and biomarkers, which directly measure changes in the brain and AD pathology to study the effects of TBI and PTSD. This proposed study will provide novel data to test these hypotheses. The results will have major implications for identifying, subjects at increased risk for AD, a possible need for early detection of AD in military Veterans with histories of TBI and PTSD, and a possible need to employ prevention and treatment measures to avoid accelerated development of AD in US military Veterans. This study is a first step toward a larger, more comprehensive study of dementia risk factors in Veterans. The results will lead to a design and statistical powering of a prevention trial. Therefore, this project could be the first step toward the prevention of AD in Veterans, and in the general population.

ELIGIBILITY:
Participants will be classified as either controls, TBI, or PTSD. General Inclusion/Exclusion Criteria will apply to all groups, with specific criteria for each group as described below.

Inclusion Criteria:

General (applies to each cohort):

* Subjects must be Veterans of the Vietnam War, 50-90 years of age. (Subjects 60-80 years of age will be selected first, while subjects <60 or >80 years of age will be added if recruitment numbers are too low in the 60-80 age range);
* Must live within 150 miles of the closest ADNI clinic in subject's area.

Specific Inclusion Criteria for Controls:

* Comparable in age, gender, and education with TBI and PTSD groups;
* May be receiving Veterans Affairs (VA) disability payments for something other than TBI or PTSD - or no disability at all.

Specific Inclusion Criteria for TBI:

* Subjects must have a documented history of moderate-severe non-penetrating TBI, which occurred during military service in Vietnam (identified from the Department of Defense or VA records);
* TBI will be defined as:

  * Loss of consciousness,
  * Post-traumatic amnesia >24 hours, OR
  * Alteration of consciousness or mental state >24 hours

Specific Inclusion Criteria for PTSD:

* Subjects who meet the Structured Clinical Interview 1 of the Diagnositic and Statistical Manual of Mental Disorders, Version IV, (Axis 1) - Text Revision [SCID-I of the DSM-IV-TR] criteria for current/chronic PTSD (identified by records, and verified by our telephone assessments);
* In addition to meeting DSM-IV-TR criteria for current/chronic PTSD, subjects must have a minimum current Clinician Administered PTSD Scale (CAPS) score of 50 as determined by telephone assessment;
* The PTSD symptoms contributing to the PTSD Diagnosis and Current CAPS score must be related to a Vietnam War related trauma.

Exclusion Criteria:

General (applies to each cohort):

* MCI/dementia;
* History of psychosis or bipolar affective disorder;
* History of alcohol or substance abuse/dependence within the past 5 years (by DSM-IV-TR criteria) or a prior prolonged history of abuse;
* MRI-related exclusions: aneurysm clips, metal implants that are determined to be unsafe for MRI; and/or claustrophobia;
* Contraindications for lumbar puncture, PET scan, or other procedures in this study;
* Any major medical condition must be stable for at least 4 months prior to enrollment. These include but are not limited to clinically significant hepatic, renal, pulmonary, metabolic or endocrine disease, cancer, HIV infection and AIDS, as well as cardiovascular disease, including:

  * cardiac surgery or myocardial infarction within the last 4 weeks;
  * unstable angina;
  * acute decompensated congestive heart failure or class IV heart failures;
  * current significant cardiac arrhythmia or conduction disturbance particularly those resulting in ventricular fibrillation, or causing syncope, or near syncope;
  * Uncontrolled high blood pressure
* Seizure disorder or any systemic illness affecting brain function during the past 5 years will be exclusionary;
* Clinical evidence of stroke;
* Have a history of relevant severe drug allergy or hypersensitivity;
* Subjects with current clinically significant unstable medical comorbidities, as indicated by history or physical exam, that pose a potential safety risk to the subject.

Specific Exclusion Criteria for Controls:

• Exclusionary criteria applied to TBI/PTSD (outlined below) will be applied to controls.

Specific Exclusion Criteria for TBI:

• Presence of PTSD by SCID-I for DSM-IV-TR criteria, or a CAPS score of >30 (Both current and/or a history of PTSD will be excluded).

Specific Exclusion Criteria for PTSD:

* Documented or self report history of mild/moderate severe TBI;
* Any history of head trauma associated with injury onset cognitive complaints; or
* Loss of consciousness for >5 minutes.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vietnam Veterans
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-10; Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Rates of change in brain regions based on neuroimaging | 1 year
  Rates of change in brain regions based on neuroimaging (magnetic resonance imaging [MRI] and amyloid positron-emission tomography [PET]) to show that those with TBI and/or PTSD have increased evidence for AD compared to Veteran controls
Rates of change in CSF amyloid beta and CSF tau/P tau levels based on biomarkers | 1 year
  Rates of change in CSF amyloid beta and CSF tau/P tau levels based on biomarkers such as cerebrospinal fluid (CSF) to show that those with TBI and/or PTSD have increased evidence for AD compared to Veteran controls
Rates of change in neuropsychological measures of memory and general cognitive performance | 1 Year
  Rates of change in neuropsychological measures of memory and general cognitive performance based on cognitive measures to show that those with TBI and/or PTSD have increased evidence for AD compared to Veteran controls

SECONDARY OUTCOMES:
Correlations within each group (TBI and PTSD) to assess whether baseline levels or rates of atrophy or cognitive decline are associated with severity of TBI or PTSD | 1 year
Group differences in the patterns of amyloid deposition (from Florbetapir F 18) and brain atrophy | 1 year
  Group differences may give insight into whether TBI or PTSD is associated with reduced brain reserve causing greater cognitive impairments as indicated by neuropsychological test performance.
Group differences in white matter integrity as assessed with Diffusion Tension Imaging (DTI) | 1 year
  Group differences in axonal damage as indicated by white matter integrity measured with DTI to determine if axonal injury resulting from TBI is associated with greater amyloid accumulation or whether brain regions with axonal damage have less amyloid accumulation due to disconnection and reduced brain activity.
Rate of change of tau deposition as measured by 18F-AV-1451 | 1 year
  Rates of change in brain regions based on Tau PET neuroimaging to show that those with TBI and/or PTSD have increased evidence for AD compared to Veteran controls

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Weiner, MD, Study Director — University of California, San Francisco; Paul Aisen, MD, Principal Investigator — USC Alzheimer's Therapeutic Research Institute (ATRI); Ronald Petersen, MD, PhD, Principal Investigator — Mayo Clinic
Locations (19):
- United States (19):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - VA Palo Alto HSC / Stanford School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Wien Center for Clinical Research, Miami Beach, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cornell Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Roper St Francis Healthcare, Charleston, South Carolina
  - U of WA / VA Puget Sound Alzheimer's Disease Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Mueller SG, Weiner MW, Thal LJ, Petersen RC, Jack CR, Jagust W, Trojanowski JQ, Toga AW, Beckett L. Ways toward an early diagnosis in Alzheimer's disease: the Alzheimer's Disease Neuroimaging Initiative (ADNI). Alzheimers Dement. 2005 Jul;1(1):55-66. doi: 10.1016/j.jalz.2005.06.003. PMID 17476317
- [Background] Weiner MW, Aisen PS, Jack CR Jr, Jagust WJ, Trojanowski JQ, Shaw L, Saykin AJ, Morris JC, Cairns N, Beckett LA, Toga A, Green R, Walter S, Soares H, Snyder P, Siemers E, Potter W, Cole PE, Schmidt M; Alzheimer's Disease Neuroimaging Initiative. The Alzheimer's disease neuroimaging initiative: progress report and future plans. Alzheimers Dement. 2010 May;6(3):202-11.e7. doi: 10.1016/j.jalz.2010.03.007. PMID 20451868
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Shaw LM, Aisen PS, Weiner MW, Petersen RC, Trojanowski JQ. Hypothetical model of dynamic biomarkers of the Alzheimer's pathological cascade. Lancet Neurol. 2010 Jan;9(1):119-28. doi: 10.1016/S1474-4422(09)70299-6. PMID 20083042
- [Background] Vemuri P, Wiste HJ, Weigand SD, Shaw LM, Trojanowski JQ, Weiner MW, Knopman DS, Petersen RC, Jack CR Jr; Alzheimer's Disease Neuroimaging Initiative. MRI and CSF biomarkers in normal, MCI, and AD subjects: predicting future clinical change. Neurology. 2009 Jul 28;73(4):294-301. doi: 10.1212/WNL.0b013e3181af79fb. PMID 19636049
- See also: Alzheimer's Disease Neuroimaging Initiative (ADNI) — http://adni.loni.usc.edu/
- See also: U.S. Department of Veterans Affairs — http://www.va.gov
- See also: Laboratory of Neuro Imaging (LONI) — https://loni.usc.edu/
- See also: Alzheimer's Therapeutic Research Institute — https://keck.usc.edu/atri/research/studies/